CLINICAL TRIAL: NCT03170531
Title: A Custom-Designed MR Coil for Spine Radiotherapy Treatment Planning
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 17-267
Record Dates: First submitted 2017-05-26; First posted 2017-05-31 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2021-05

CONDITIONS: Healthy
Keywords: MRI; MR imaging; 17-267

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Custom MR spine coil
  Interventions: Diagnostic Test: Custom Designed Spine Coil; Diagnostic Test: FDA approved spine coil

INTERVENTIONS:
Diagnostic Test: Custom Designed Spine Coil — During the participant's MR scan, the custom spine coil will be placed between the participant and the immobilization mold. image parameters will be optimized for spine anatomy for the pulse sequences which are standard for MR imaging.
Diagnostic Test: FDA approved spine coil — During the participant's MR scan, the FDA spine coil will be placed between the participant and the immobilization mold. image parameters will be optimized for spine anatomy for the pulse sequences which are standard for MR imaging. Volunteers may receive up to 3 scans to allow for comparisons of changes to the calibration files as we continue to test the coil and improve its performance.

SUMMARY:
The purpose of this study is to assess the image quality improvement provided by a custom MR spine coil in comparison with the FDA approved coil when used for radiotherapy treatment planning.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Volunteers age 18 or older

Exclusion Criteria:

* Anyone who would be normally excluded from undergoing an MRI examination as per Memorial Hospital for Cancer and Allied Diseases Screening Questionnaire
* Volunteers with a pacemaker, aneurysm clip or any other condition that would warrant avoidance of a strong magnetic field
* Female volunteers who are pregnant or nursing
* Volunteers who are unable to comply or complete the MRI exam due to claustrophobia or high levels of anxiety
* Volunteers who are under direct supervision of any investigators on the study will not be eligible to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Enrollment in this study will be open to all MSKCC employees to act as healthy volunteers provided they meet the eligibility criteria for the protocol. Employees who provide consent willfully and voluntarily may participate as a healthy volunteer once. Employees who are under direct supervision of any investigators on the study will not be eligible to participate. An IRB approved flyer with pertinent contact information will be distributed throughout the institution to inform all MSKCC employees of the possibility of participating in this study. No preferences will be given by race or gender for the selection of participants.
Sampling Method: Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2017-05-23 (Actual); Primary Completion 2021-04-26 (Actual); Study Completion 2021-04-26 (Actual)

PRIMARY OUTCOMES:
Optimize performance | Day of intervention
  Optimize performance of custom-designed spine coil in RT configuration on participants. This objective focuses on the technology of the custom designed spine coil and does not require any statistical analysis.
Compare the signal-to-noise ratio of a custom spine coil with the existing FDA approved posterior coil array used for spine imaging | Day of intervention
  To quantify image quality obtained from the custom spine coil and the existing coil, SNR will be calculated (see Section 4.1 for details) for both coils. If, for a volunteer, the SNR from the custom coil is larger than 105% of that from the existing coil (we insist a 5% improvement margin due to anticipated uncertainty and variability), then we will classify this sample point as a "success". We will combine the 15 volunteers from the three cohorts (cervical-spine, thoracic-spine and lumbar-spine) and impose the following decision rule: If at least 12 out of the total 15 volunteers are success, then we declare the custom designed spine coil promising and worthy of further investigation.

CONTACTS AND LOCATIONS:
Locations (1):
- Memorial Sloan - Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://mskcc.org